CLINICAL TRIAL: NCT02614183
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 in Patients With Episodic Migraine - the EVOLVE-1 Study
Brief Title: Evaluation of Galcanezumab in the Prevention of Episodic Migraine- the EVOLVE-1 Study
Acronym: EVOLVE-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15767; I5Q-MC-CGAG (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Migraine
Keywords: prevention; prophylaxis; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Galcanezumab 120mg (Experimental): Galcanezumab given by subcutaneous (SC) injection at 120mg dose once a month for 6 months. Participants received a loading dose of 240mg (2 injections of 120mg each) was administered at visit 3 only.
  Interventions: Drug: Galcanezumab
- Galcanezumab 240mg (Experimental): Galcanezumab 240mg given by SC injection once a month for 6 months.
  Interventions: Drug: Galcanezumab
- Placebo (Placebo Comparator): Placebo given by SC injection once a month for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742
  Arms: Galcanezumab 120mg; Galcanezumab 240mg
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of the study drug known as galcanezumab in participants with episodic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of episodic migraine as defined by International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 beta guidelines (1.1 or 1.2) (ICHD-3 2013), with a history of migraine headaches of at least 1 year prior to screening, migraine onset prior to age 50 and MONTHLY frequency of 4-14 Migraine Headache Days (MHD).

Exclusion Criteria:

* Are currently enrolled in or have participated within the last 30 days or within 5 half-lives (whichever is longer) in a clinical trial involving an investigational product.
* Current use or prior exposure to Galcanezumab or another CGRP antibody.
* Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins, or to Galcanezumab.
* History of persistent daily headache, cluster headache or migraine subtypes including hemiplegic (sporadic or familial) migraine, ophthalmoplegic migraine, and migraine with brainstem aura (basilar-type migraine) defined by IHS ICHD-3 beta.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 862 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (95):
- United States (80):
  - Territory Neurology & Research Institute, Tucson, Arizona
  - Orange Grove Family Practice, Tucson, Arizona
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Advanced Clinical Research, Carmichael, California
  - Pharmacology Research Institute, Newport Beach, Encino, California
  - Tooraj Joseph Raoof M.D., Inc., Encino, California
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Sun Valley Research Center, Imperial, California
  - Irvine Clinical Research Center, Irvine, California
  - Pharmacology Research Institute, Newport Beach, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, Newport Beach, California
  - Desert Valley Research, Rancho Mirage, California
  - Anderson Clinical Research, Redlands, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Mile High Research Center, Denver, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - Advanced Neurosciences Research, LLC, Fort Collins, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Meridien Research, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Psychiatric Inst of Florida-Clinical Neuroscience Solutions, Orlando, Florida
  - Compass Research, Oviedo, Florida
  - Accord Clinical Research, LLC, Port Orange, Florida
  - Roskamp Institute, Sarasota, Florida
  - Infinity Clinical Reserach . LLC, Sunrise, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Advanced Clinical Research LLC, Meridian, Idaho
  - Healthcare Research Network - Blue Island, Blue Island, Illinois
  - Community Clinical Research Center, Anderson, Indiana
  - Investigative Clinical Research of Indiana, LLC, Elwood, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Deaconess Clinic Inc, Newburgh, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Phoenix Medical Research, Inc, Prairie Village, Kansas
  - Otri-Med Corporation, Edgewood, Kentucky
  - L-Marc Research Center, Louisville, Kentucky
  - PharmaSite Research Inc, Baltimore, Maryland
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - Michigan Head, Pain and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - ClinVest, Springfield, Missouri
  - Healthy Perspectives Innovative Mental Health Services, PL, Nashua, New Hampshire
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Dent Neurological Institute, Amherst, New York
  - Central New York Clinical Research, Manlius, New York
  - NYU Langone, New York, New York
  - Fieve Clincial Services, New York, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Metrolina Neurological Associates, PA, Charlotte, North Carolina
  - Headache Wellness Center, Greensboro, North Carolina
  - Rapid Medical Research Inc, Cleveland, Ohio
  - Medical College of Ohio at Toledo, Toledo, Ohio
  - Healthcare Research Consultant, Tulsa, Oklahoma
  - Summit Research Network Inc, Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - 8 Medical Park, Columbia, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Clinical Research Associates, Nashville, Tennessee
  - FutureSearch Trials, Austin, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Radiant Research - San Antonio, San Antonio, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - National Clinical Research - Richmond, Richmond, Virginia
  - Premier Clinical Research, Spokane, Washington
  - Vancouver Clinic, Vancouver, Washington
  - Clinical Investigation Specialists Inc, Kenosha, Wisconsin
- Canada (9):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Brampton
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Kelowna
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Mississauga
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ottawa
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Sherbrooke
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Toronto
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Vancouver
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Waterloo
- Puerto Rico (6):
  - Office of Dr. Ruddy Guerra, Manatí
  - NuFrontiers Clinical Research LLC, Rio Piedras
  - Clinical Research Puerto Rico, Inc., San Juan
  - GCM Medical Group PSC, San Juan
  - Instituto de Neurologia Dra. Ivonne Fraga, San Juan
  - Neuro GI Wellness Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Ailani J, Kuruppu DK, Rettiganti M, Oakes T, Schroeder K, Wietecha L, Port M, Blumenfeld AM. Does "wearing off" of efficacy occur in galcanezumab-treated patients at the end of the monthly treatment cycle? Post hoc analyses of four phase III randomized trials. Headache. 2022 Feb;62(2):198-207. doi: 10.1111/head.14257. Epub 2022 Jan 25. PMID 35076090
- [Derived] Citrome L, Sanchez Del Rio M, Dong Y, Nichols RM, Tockhorn-Heidenreich A, Foster SA, Stauffer VL. Benefit-Risk Assessment of Galcanezumab Versus Placebo for the Treatment of Episodic and Chronic Migraine Using the Metrics of Number Needed to Treat and Number Needed to Harm. Adv Ther. 2021 Aug;38(8):4442-4460. doi: 10.1007/s12325-021-01848-x. Epub 2021 Jul 15. PMID 34264500
- [Derived] Jedynak J, Eross E, Gendolla A, Rettiganti M, Stauffer VL. Shift from high-frequency to low-frequency episodic migraine in patients treated with Galcanezumab: results from two global randomized clinical trials. J Headache Pain. 2021 May 28;22(1):48. doi: 10.1186/s10194-021-01222-w. PMID 34049484
- [Derived] Pozo-Rosich P, Samaan KH, Schwedt TJ, Nicholson RA, Rettiganti M, Pearlman EM. Galcanezumab Provides Consistent Efficacy Throughout the Dosing Interval Among Patients with Episodic and Chronic Migraine: A Post Hoc Analysis. Adv Ther. 2021 Jun;38(6):3154-3165. doi: 10.1007/s12325-021-01708-8. Epub 2021 May 5. PMID 33950375
- [Derived] Ament M, Day K, Stauffer VL, Skljarevski V, Rettiganti M, Pearlman E, Aurora SK. Effect of galcanezumab on severity and symptoms of migraine in phase 3 trials in patients with episodic or chronic migraine. J Headache Pain. 2021 Feb 6;22(1):6. doi: 10.1186/s10194-021-01215-9. PMID 33549036
- [Derived] Kuruppu DK, North JM, Kovacik AJ, Dong Y, Pearlman EM, Hutchinson SL. Onset, Maintenance, and Cessation of Effect of Galcanezumab for Prevention of Migraine: A Narrative Review of Three Randomized Placebo-Controlled Trials. Adv Ther. 2021 Mar;38(3):1614-1626. doi: 10.1007/s12325-021-01632-x. Epub 2021 Feb 5. PMID 33544305
- [Derived] Dodick DW, Doty EG, Aurora SK, Ruff DD, Stauffer VL, Jedynak J, Dong Y, Pearlman EM. Medication overuse in a subgroup analysis of phase 3 placebo-controlled studies of galcanezumab in the prevention of episodic and chronic migraine. Cephalalgia. 2021 Mar;41(3):340-352. doi: 10.1177/0333102420966658. Epub 2020 Nov 3. PMID 33143451
- [Derived] Ailani J, Andrews JS, Rettiganti M, Nicholson RA. Impact of galcanezumab on total pain burden: findings from phase 3 randomized, double-blind, placebo-controlled studies in patients with episodic or chronic migraine (EVOLVE-1, EVOLVE-2, and REGAIN trials). J Headache Pain. 2020 Oct 17;21(1):123. doi: 10.1186/s10194-020-01190-7. PMID 33069214
- [Derived] Stauffer VL, Turner I, Kemmer P, Kielbasa W, Day K, Port M, Quinlan T, Camporeale A. Effect of age on pharmacokinetics, efficacy, and safety of galcanezumab treatment in adult patients with migraine: results from six phase 2 and phase 3 randomized clinical trials. J Headache Pain. 2020 Jun 23;21(1):79. doi: 10.1186/s10194-020-01148-9. PMID 32576229
- [Derived] Bangs ME, Kudrow D, Wang S, Oakes TM, Terwindt GM, Magis D, Yunes-Medina L, Stauffer VL. Safety and tolerability of monthly galcanezumab injections in patients with migraine: integrated results from migraine clinical studies. BMC Neurol. 2020 Jan 17;20(1):25. doi: 10.1186/s12883-020-1609-7. PMID 31952501
- [Derived] Kielbasa W, Quinlan T. Population Pharmacokinetics of Galcanezumab, an Anti-CGRP Antibody, Following Subcutaneous Dosing to Healthy Individuals and Patients With Migraine. J Clin Pharmacol. 2020 Feb;60(2):229-239. doi: 10.1002/jcph.1511. Epub 2019 Sep 4. PMID 31482569
- [Derived] Silberstein SD, Stauffer VL, Day KA, Lipsius S, Wilson MC. Galcanezumab in episodic migraine: subgroup analyses of efficacy by high versus low frequency of migraine headaches in phase 3 studies (EVOLVE-1 & EVOLVE-2). J Headache Pain. 2019 Jun 28;20(1):75. doi: 10.1186/s10194-019-1024-x. PMID 31253091
- [Derived] Stauffer VL, Wang S, Voulgaropoulos M, Skljarevski V, Kovacik A, Aurora SK. Effect of Galcanezumab Following Treatment Cessation in Patients With Migraine: Results From 2 Randomized Phase 3 Trials. Headache. 2019 Jun;59(6):834-847. doi: 10.1111/head.13508. Epub 2019 Apr 3. PMID 30942898
- [Derived] Forderreuther S, Zhang Q, Stauffer VL, Aurora SK, Lainez MJA. Preventive effects of galcanezumab in adult patients with episodic or chronic migraine are persistent: data from the phase 3, randomized, double-blind, placebo-controlled EVOLVE-1, EVOLVE-2, and REGAIN studies. J Headache Pain. 2018 Dec 29;19(1):121. doi: 10.1186/s10194-018-0951-2. PMID 30594122
- [Derived] Nichols R, Doty E, Sacco S, Ruff D, Pearlman E, Aurora SK. Analysis of Initial Nonresponders to Galcanezumab in Patients With Episodic or Chronic Migraine: Results From the EVOLVE-1, EVOLVE-2, and REGAIN Randomized, Double-Blind, Placebo-Controlled Studies. Headache. 2019 Feb;59(2):192-204. doi: 10.1111/head.13443. Epub 2018 Nov 21. PMID 30462830
- [Derived] Stauffer VL, Dodick DW, Zhang Q, Carter JN, Ailani J, Conley RR. Evaluation of Galcanezumab for the Prevention of Episodic Migraine: The EVOLVE-1 Randomized Clinical Trial. JAMA Neurol. 2018 Sep 1;75(9):1080-1088. doi: 10.1001/jamaneurol.2018.1212. PMID 29813147
- See also: Click here for more information about this study: Evaluation of Galcanezumab in the Prevention of Episodic Migraine- the EVOLVE-1 Study — http://www.lillytrialguide.com/EN-us/studies/headache/cgag

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants (pts) received placebo by subcutaneous injection once a month for 6 months. Participants did not receive any intervention during post-treatment follow-up phase.
- Galcanezumab 120mg: Participants received loading dose of 240mg (2 injections of 120mg each) galcanezumab at first doing visit followed by 120mg galcanezumab once a month for 5 months by subcutaneous injection. Participants did not receive any intervention during post-treatment follow-up phase.
- Galcanezumab 240mg: Participants received 240mg galcanezumab by subcutaneous injection once a month for 6 months. Participants did not receive any intervention during post-treatment follow-up phase.
Period: Double Blind Treatment Phase
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Started | 434 | 214 | 214
Received at Least One Dose of Study Drug | 433 | 213 | 212
Safety Population | 432 | 206 (One pt randomized to placebo received galcanezumab 120mg due to dosing error moved to this group.) | 220 (Eight pts discontinued after loading dose of 240mg galcanezumab in 120mg group moved to this group.)
Completed | 351 | 177 | 175
Not Completed | 83 | 37 | 39
Not completed — Adverse Event | 10 | 9 | 7
Not completed — Lack of Efficacy | 10 | 1 | 2
Not completed — Lost to Follow-up | 18 | 9 | 5
Not completed — Physician Decision | 7 | 3 | 2
Not completed — Pregnancy | 2 | 1 | 3
Not completed — Protocol Violation | 2 | 2 | 2
Not completed — Withdrawal by Subject | 33 | 11 | 16
Not completed — Did not receive study drug | 1 | 1 | 2
Period: Post Treatment Follow-up Phase
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Started | 372 (Participants who discontinued double blind phase had an option to enter post-treatment phase.) | 185 (Participants who discontinued double blind phase had an option to enter post-treatment phase.) | 183 (Participants who discontinued double blind phase had an option to enter post-treatment phase.)
Safety Population | 372 | 183 | 185 (Two participants who received only 240mg loading dose prior to discontinuation moved to this group.)
Completed | 354 | 179 | 171
Not Completed | 18 | 6 | 12
Not completed — Lost to Follow-up | 5 | 3 | 5
Not completed — Physician Decision | 5 | 1 | 2
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 2 | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received placebo by subcutaneous injection once a month for 6 months. Participants did not receive any intervention during post-treatment follow-up phase.
- Total: Total of all reporting groups
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg | Total
Number analyzed (Participants) | 433 | 213 | 212 | 858
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.33 (11.40) | 40.93 (11.87) | 39.07 (11.52) | 40.67 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 362 | 181 | 175 | 718
  Male | 71 | 32 | 37 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 58 | 27 | 37 | 122
  Not Hispanic or Latino | 359 | 180 | 171 | 710
  Unknown or Not Reported | 16 | 6 | 4 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 3 | 3
  Asian | 13 | 7 | 4 | 24
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 3
  Black or African American | 42 | 29 | 23 | 94
  White | 356 | 169 | 165 | 690
  More than one race | 21 | 8 | 15 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 44 | 20 | 21 | 85
  Puerto Rico | 11 | 5 | 4 | 20
  United States | 378 | 188 | 187 | 753
Migraine Headache Days (MHD) per month [Mean (Standard Deviation); unit: Days per Month] — Migraine Headache Day (MHD): A calendar day on which a migraine headache or probable migraine headache occurred.
  Days per Month | 9.08 (2.97) | 9.21 (3.05) | 9.14 (2.91) | 9.13 (2.97)

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days
Description: Migraine Headache Day (MHD):A calendar day on which a migraine headache or probable migraine headache occurred.
  Migraine Headache : A headache, with or without aura, of ≥30 minutes duration with both of the following required features (A and B):
  A) At least 2 of the following headache characteristics: Unilateral location; Pulsatile quality; Moderate or severe pain intensity; Aggravation by or causing avoidance of routine physical activity; AND B) During headache at least one of the following: Nausea and/or vomiting; Photophobia and phonophobia;
  Overall mean is derived from the average of months 1 to 6 from mixed model repeated measures (MMRM) model. Least Square (LS) mean was calculated using mixed model repeated measures (MMRM) model with treatment, pooled country, month, and treatment by month, baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 6
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline value.
Measure: Least Squares Mean (Standard Error); unit: Days
Groups:
- Placebo: Participants received placebo by subcutaneous injection once a month for 6 months.
- Galcanezumab 120mg: Participants received loading dose of 240mg (2 injections of 120mg each) galcanezumab at first doing visit followed by 120mg galcanezumab once a month for 5 months by subcutaneous injection.
- Galcanezumab 240mg: Participants received 240mg galcanezumab by subcutaneous injection once a month for 6 months.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 425 | 210 | 208
Days | -2.81 (0.24) | -4.73 (0.29) | -4.57 (0.29)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -1.92, 95% CI 2-sided [-2.48 to -1.37], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-2.31 to -1.20], Standard Error of Mean 0.28

2. Secondary Outcome: Mean Percentage of Participants With Reduction From Baseline ≥50%, ≥75% and 100% in Monthly Migraine Headache Days
Description: Migraine Headache Day (MHD): A calendar day on which a migraine headache or probable migraine headache occurred.
  Mean is derived from the average of months 1 to 6 from generalized linear mixed model repeated measures. Mean percentages of participants were calculated with a generalized linear mixed model repeated measures method with treatment, month and treatment by month, baseline.
Time Frame: Baseline, Month 1 through Month 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 425 | 210 | 208
percentage of participants
  ≥50% | 38.6 (1.7) | 62.3 (2.4) | 60.9 (2.5)
  ≥75% | 19.3 (1.4) | 38.8 (2.4) | 38.5 (2.4)
  100% | 6.2 (0.8) | 15.6 (1.6) | 14.6 (1.6)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Reduction from Baseline ≥50%; Test type: Superiority; Odds Ratio (OR) = 2.63, 95% CI 2-sided [2.05 to 3.37]
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Reduction from Baseline ≥50%; Test type: Superiority; Odds Ratio (OR) = 2.48, 95% CI 2-sided [1.94 to 3.18]
Statistical Analysis 3: Comparison: Placebo vs Galcanezumab 120mg; Reduction from Baseline ≥75%; Test type: Superiority; Odds Ratio (OR) = 2.65, 95% CI 2-sided [2.04 to 3.45]
Statistical Analysis 4: Comparison: Placebo vs Galcanezumab 240mg; Reduction from Baseline ≥75%; Test type: Superiority; Odds Ratio (OR) = 2.62, 95% CI 2-sided [2.01 to 3.41]
Statistical Analysis 5: Comparison: Placebo vs Galcanezumab 120mg; Reduction from Baseline = 100%; Test type: Superiority; Odds Ratio (OR) = 2.80, 95% CI 2-sided [1.96 to 4.01]
Statistical Analysis 6: Comparison: Placebo vs Galcanezumab 240mg; Reduction from Baseline = 100%; Test type: Superiority; Odds Ratio (OR) = 2.61, 95% CI 2-sided [1.81 to 3.75]

3. Secondary Outcome: Mean Change From Baseline in the Migraine-Specific Quality of Life Questionnaire (MSQ) Version 2.1 (v2.1) Role Function Restrictive Domain
Description: MSQ v2.1 was developed to address physical & emotional limitations of specific concern to individuals with migraine.
  It consists of 14 items that address 3 domains:(1) Role Function-Restrictive (items 1-7);(2) Role Function- Preventive (items 8-11);&(3) Emotional Function (items 12-14).Response options range from "none of the time" (value 1) to "all of the time" (value 6), & are reverse-recoded (value 6 to 1) before the domain scores are calculated.Total raw scores for each domain is the sum of the final item value for all of the items in that domain.After the total raw score is computed for each domain, they are transformed to a 0-100 scale with higher scores indicating a better health status & a positive change in scores reflecting functional improvement.
  Mean is derived from the average of months 4 to 6 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline by month & baseline MHD category as fixed factors.
Time Frame: Baseline, Month 4 through Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 419 | 207 | 202
units on a scale | 24.69 (1.07) | 32.43 (1.31) | 32.09 (1.32)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = 7.74, 95% CI 2-sided [5.20 to 10.28], Standard Error of Mean 1.29
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = 7.40, 95% CI 2-sided [4.83 to 9.97], Standard Error of Mean 1.31

4. Secondary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days Requiring Medication for the Acute Treatment of Migraine or Headache
Description: Migraine Headache Day (MHD):A calendar day on which a migraine headache or probable migraine headache occurred.
  Overall mean is derived from the average of months 1 to 6 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, baseline by month, and baseline MHD category as fixed effects.
Time Frame: Baseline, Month 1 through Month 6
Population: All randomized participants who received at least one dose of study drug and had baseline and post baseline value.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 425 | 210 | 208
Days | -2.15 (0.21) | -3.96 (0.25) | -3.76 (0.26)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-2.28 to -1.33], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; Odds Ratio (OR) = -1.61, 95% CI 2-sided [-2.09 to -1.14], Standard Error of Mean 0.26

5. Secondary Outcome: Mean Change From Baseline in the Patient Global Impression of Severity (PGI-S) Rating
Description: The PGI-S scale is a patient-rated instrument that measures patients own global impression of their illness severity. The patient was instructed as follows: "Considering migraine as a chronic condition, how would you rate your level of illness?" Response options were from 1 ("normal, not at all ill") to 7 ("extremely ill"). Mean is derived from the average of months 4 to 6 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, baseline by month, and baseline MHD category as fixed factors.
Time Frame: Baseline, Month 4 through Month 6
Population: All randomized participants who received at least one dose of study drug and had baseline and post baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 419 | 207 | 202
units on a scale | -1.27 (0.08) | -1.59 (0.10) | -1.55 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.52 to -0.12], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.48 to -0.07], Standard Error of Mean 0.10

6. Secondary Outcome: Overall Mean Change From Baseline in Headache Hours
Description: Headache Hours is calculated as the total number of headache hours on which a headache occurred. Overall mean is derived from the average of months 1 to 6 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, baseline by month and baseline MHD category.
Time Frame: Baseline, Month 1 through Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Hours per Month
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 425 | 210 | 208
Hours per Month | -15.67 (2.24) | -29.65 (2.70) | -29.31 (2.72)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -13.98, 95% CI 2-sided [-18.99 to -8.97], Standard Error of Mean 2.55
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -13.64, 95% CI 2-sided [-18.68 to -8.60], Standard Error of Mean 2.57

7. Secondary Outcome: Mean Change From Baseline on the Migraine Disability Assessment Test (MIDAS) Total Score
Description: The MIDAS is a participant-rated scale which was designed to quantify headache-related disability over a 3-month period. This instrument consists of five items that reflect the number of days reported as missing or with reduced productivity at work or home, and the number of days of missed social events. Each item has a numeric response range from 0 to 90 days, if days are missed from work or home they are not counted as days with reduced productivity at work or home. The numeric responses are summed to produce a total score ranging from 0 to 270, in which a higher value is indicative of more disability.
  LSMean was calculated using MMRM model with treatment, pooled country, month, treatment by month, baseline, baseline by month, and baseline MHD category as fixed factors.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 389 | 195 | 189
units on a scale | -14.87 (1.37) | -21.16 (1.65) | -20.06 (1.68)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -6.29, 95% CI 2-sided [-9.45 to -3.13], Standard Error of Mean 1.61
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; Mean Difference (Final Values) = -5.19, 95% CI 2-sided [-8.39 to -1.98], Standard Error of Mean 1.63

8. Secondary Outcome: Percentage of Participants Developing Anti-drug Antibodies (ADA) to Galcanezumab
Description: Treatment emergent (TE) ADA evaluable participant is considered to be TE ADA+ if the subject has at least one post-baseline titer that is a 4-fold or greater increase in titer from baseline measurement. If baseline result is ADA Not Present, then the participant is TE ADA+ if there is at least one post-baseline result of ADA present with titer >= 1: 20.
Time Frame: Month 1 through Month 6
Population: All randomized participants who received at least one dose of study drug and had least one non-missing test result for ADA for each of the baseline period and the post-baseline period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 422 | 202 | 213
percentage of participants
  TE ADA+ | 1.66 | 3.47 | 5.16
  Neutralizing Antibodies | 1.42 | 3.47 | 5.16
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; TE ADA Positive; Test type: Superiority; p < .160, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; TE ADA Positive; Test type: Superiority; p = .020, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs Galcanezumab 120mg; Neutralizing Antibodies; Test type: Superiority; p = .131, Fisher Exact
Statistical Analysis 4: Comparison: Placebo vs Galcanezumab 240mg; Neutralizing Antibodies; Test type: Superiority; p = .009, Fisher Exact

9. Secondary Outcome: Pharmacokinetics (PK): Serum Concentrations of Galcanezumab
Description: Pharmacokinetics (PK): Serum Concentrations of Galcanezumab.
Time Frame: Month 6
Population: All randomized participants who received at least one dose of study drug and had measurable serum concentrations.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 156 | 149
Nanogram per milliliter (ng/mL) | 15400 (8340) | 29500 (12300)

10. Secondary Outcome: Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP)
Description: Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP).
Time Frame: Month 6
Population: All randomized participants who had received at least one dose of study drug and had measurable plasma concentrations.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 28 | 165 | 158
ng/mL | 0.888 (1.89) | 4.25 (1.79) | 5.13 (2.43)

ADVERSE EVENTS:
Time Frame: Up to 10 Months
Description: All-Cause Mortality:All participants (pts) who received atleast 1 dose of study drug.
  SAE/AE:Eight pts discontinued after receiving loading dose (LD) of 240mg galcanezumab (GAL) in 120mg group (gp) moved to 240mg treatment gp. One pt randomized to placebo received GAL 120mg due to dosing error moved to 120mg treatment gp. Two pts who received only 240mg LD prior to discontinuation moved to 240mg post-treatment gp. There are gender specific adverse events only occurring in male or female pts.
Groups:
- Placebo - Treatment Phase: Participants received placebo by subcutaneous injection once a month for 6 months.
- Galcanezumab 120mg - Treatment Phase: Participants received loading dose of 240mg (2 injections of 120mg each) galcanezumab at first doing visit followed by 120mg galcanezumab once a month for 5 months by subcutaneous injection.
- Galcanezumab 240mg - Treatment Phase: Participants received 240mg galcanezumab by subcutaneous injection once a month for 6 months.
- Placebo - Post-Treatment Phase; Galcanezumab 120mg - Post-Treatment Phase; Galcanezumab 240mg - Post-Treatment Phase: Participants didn't receive any intervention.
Arm/Group | Placebo - Treatment Phase | Galcanezumab 120mg - Treatment Phase | Galcanezumab 240mg - Treatment Phase | Placebo - Post-Treatment Phase | Galcanezumab 120mg - Post-Treatment Phase | Galcanezumab 240mg - Post-Treatment Phase
All-Cause Mortality (participants affected / at risk) | 0/433 | 0/213 | 0/212 | 0/372 | 0/185 | 0/183
Serious Adverse Events (participants affected / at risk) | 5/432 | 6/206 | 0/220 | 2/372 | 4/183 | 4/185
Other Adverse Events (participants affected / at risk) | 129/432 | 63/206 | 72/220 | 22/372 | 12/183 | 12/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Treatment Phase (N=432) | Galcanezumab 120mg - Treatment Phase (N=206) | Galcanezumab 240mg - Treatment Phase (N=220) | Placebo - Post-Treatment Phase (N=372) | Galcanezumab 120mg - Post-Treatment Phase (N=183) | Galcanezumab 240mg - Post-Treatment Phase (N=185)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tubular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/361 (0) | 0/175 (0) | 0/182 (0) | 0/311 (0) | 1/156 (1) | 0/156 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0/361 (0) | 0/175 (0) | 0/182 (0) | 0/311 (0) | 0/156 (0) | 1/156 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0/361 (0) | 0/175 (0) | 0/182 (0) | 0/311 (0) | 1/156 (1) | 0/156 (0)
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Treatment Phase (N=432) | Galcanezumab 120mg - Treatment Phase (N=206) | Galcanezumab 240mg - Treatment Phase (N=220) | Placebo - Post-Treatment Phase (N=372) | Galcanezumab 120mg - Post-Treatment Phase (N=183) | Galcanezumab 240mg - Post-Treatment Phase (N=185)
Injection site pain (General disorders) | 75 (365) | 33 (158) | 45 (212) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 4 (11) | 7 (14) | 12 (20) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 31 (36) | 9 (11) | 15 (18) | 12 (14) | 6 (6) | 5 (5)
Urinary tract infection (Infections and infestations) | 15 (15) | 8 (9) | 13 (13) | 8 (8) | 3 (3) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 29 (31) | 19 (23) | 8 (9) | 3 (3) | 3 (3) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-09-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT02614183/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT02614183/SAP_001.pdf